CLINICAL TRIAL: NCT06164431
Title: Single-dose, Open-label, Randomized, Crossover Bioavailability Study of 200mg Tablets ZSP1273 Versus 200mg Granules ZSP1273 Under Fasted Condition in Healthy Participants
Brief Title: Bioavailability Study in Healthy Participants, 200mg Tablets ZSP1273 Versus 200mg Granules ZSP1273
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ZSP1273-22-09
Record Dates: First submitted 2023-11-30; First posted 2023-12-11 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Bioequivalence
MeSH Terms: interventions — ZSP1273

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZSP1273 Sequence 1 (Experimental): Single oral dose of 200mg ZSP1273 tablet administered under fasting conditions in first period and 200mg granules in second period，then 200mg ZSP1273 tablet administered under fasting conditions in third period and 200mg granules in fourth period.
  Interventions: Drug: ZSP1273 tablet; Drug: zsp1273 granules
- ZSP1273 Sequence 2 (Experimental): Single oral dose of 200mg ZSP1273 granules administered under fasting conditions in first period and 200mg tablet in second period，then 200mg ZSP1273 granules administered under fasting conditions in third period and 200mg tablet in fourth period.
  Interventions: Drug: ZSP1273 tablet; Drug: zsp1273 granules

INTERVENTIONS:
Drug: ZSP1273 tablet — Participants receive ZSP1273 tablet orally.
Drug: zsp1273 granules — Participants receive ZSP1273 granules orally.

SUMMARY:
The purpose of this study is to establish bioavailability of 2 treatments with ZSP1273: 200mg tablets and 200mg granules will be given to healthy Participants under fasting conditions.

Bioavailability will be evaluated and verified on the basis of pharmacokinetic data.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) ≥19 to ≤26kg/m2 and total body weight >50 kg at Screening (calculated as a function of measured height and weight according to the formula, BMI = kg / m2 where m2 is height in meters squared);
2. Ability to understand and willingness to sign a written informed consent form;
3. Normal physical examination, vital signs, 12-lead ECG, and clinical laboratory values, or any abnormality that is non-clinically significant.

Exclusion Criteria:

1. Participants with an allergic disposition (multiple drug and food allergies) or who, as determined by the investigator, are likely to be allergic to the investigational drug product or any component of the investigational drug product.
2. Participants had taken prescription, over-the-counter, herbal, or vitamin products within 14 days prior to screening；
3. Smoking more than 5 cigarettes per day within 3 months prior to screening，or who cannot stop using any tobacco products during the study period;
4. Participants who donated blood/bleeding profusely (> 400 mL) 3 months prior to randomization;
5. Those with clinically significant Electrocardiogram(ECG) abnormalities, or QTcF > 450ms;
6. Participants who test positive at screening for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), Hepatitis C virus (HCV) antibody or Syphilis spirochete-specific antibodies (TPPA);
7. Participants who test positive at Screening and/or admission (Day -1) for alcohol abuse.
8. Females who are pregnant, lactating, or likely to become pregnant during the study.
9. History of dysphagia or any gastrointestinal disorder that affect absorption

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Day 1 to Day 20
  The Cmax of a single dose of ZSP1273 tablet and ZSP1273 granules will be evaluated and compared.
Area under the concentration-time curve from time zero to infinity (AUCinf) | Day 1 to Day 20
  The AUCinf of a single dose of ZSP1273 tablet and ZSP1273 granules will be evaluated and compared.
Area under the concentration-time curve from time zero to last time of quantifiable concentration (AUClast) | Day 1 to Day 20
  The AUClast of a single dose of ZSP1273 tablet and ZSP1273 granules will be evaluated and compared.

SECONDARY OUTCOMES:
Number of participants with drug-related adverse events as assessed by CTCAE v5.0 | Day 1 to Day 20

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Hospital of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided